CLINICAL TRIAL: NCT01252810
Title: A Phase 2, Double-Blind, Randomized, Safety Study of GE-145 320 mg I/mL Injection Versus Iopamidol 370 mg I/mL in Elderly Subjects Undergoing Coronary Artery Catheterization Procedure
Brief Title: Safety Study of GE-145 320 mg I/mL Injection vs. Iopamidol 370 mg I/mL in Elderly Subjects Undergoing Coronary Procedure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: i3 Statprobe (Industry); Medpace, Inc. (Industry); Biomedical Systems (Industry); Rules-Based Medicine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: GE 145-002
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Results first posted 2014-05-02 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Chronic Renal Insufficiency; Diabete Mellitus; Congestive Heart Failure
Keywords: CATH Catheterization; CI-AKI Contrast-induced acute kidney injury; DM Diabetes mellitus; eGFR Estimated glomerular filtration rate; MDRD Modification of Diet in Renal Disease; NYHA New York Heart Association; PCI Percutaneous coronary intervention; SCr Serum creatinine
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus; Heart Failure | interventions — 5-(formyl-(3-(formyl-(3,5-bis (2,3-dihydroxypropylcarbamoyl)-2,4,6-triiodophenyl) amino)-2-hydroxypropyl)amino)-N,N'-bis(2,3-dihydroxypropyl)-2,4,6-triiodobenzene-1,3-dicarboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GE 145 320mg I/ml injection (Experimental)
  Interventions: Drug: GE-145
- Iopamidol 370mg I/ml injection (Active Comparator)
  Interventions: Drug: GE-145

INTERVENTIONS:
Drug: GE-145 — GE-145-320 mg I/mL as a single iv. administration. Comparator agent Isovue (iopamidol) 370 mg I/mL as a single iv. administration.
  Other Names: Ioforminol

SUMMARY:
To evaluate cardio-renal and overall safety profile of GE 145 320 mg I/ml Injection when compared to iopamidol 370 mg I/mL. The study will focus on elderly subjects with either chronic renal insufficiency, or diabetes mellitus (DM) requiring drug therapy, or congestive heart failure (CHF) NYHA Class III or greater, who are referred for a coronary catheterization procedure with or without PCI.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 65 years of age with cardiovascular disease who are referred for a coronary catheterization procedure with or without PCI.
* The subject has at least one of the following comorbidities:
* 1) Chronic renal insufficiency, (eGFR <60 but 15 mL/min/1.73 m2 according to the MDRD equation) as measured within 2 weeks or at the screening visit;
* 2) DM diagnosed greater than 6 months prior to study entry and which requires either insulin or anti-hyperglycemic drug therapy;
* 3) CHF (NYHA) class III or greater measured within 2 weeks of enrollment or at the screening visit.

Exclusion Criteria:

* The subject has known allergies to either iodine or any ICM.
* The subject has severe renal insufficiency (eGFR <15 mL/min/1.73 m2 according to the MDRD equation) or is on dialysis.
* The subject has acute coronary syndrome requiring emergency coronary angiography and/or intervention.
* The subject is not willing or unable to discontinue metformin (e.g., Glucophage) at the time of the study procedure.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 284 (Actual)
Dates: Start 2010-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rubin Sheng, M.D., Study Director — GE Healthcare
Locations (1):
- GE Healthcare, Princeton, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ioforminol 320mg I/ml Injection: Ioforminol 320 mg I/mL as a single iv. administration.
- Iopamidol 370mg I/ml Injection: Iopamidol 370 mg I/mL as a single iv. administration.
Period: Overall Study
Arm/Group | Ioforminol 320mg I/ml Injection | Iopamidol 370mg I/ml Injection
Started | 142 | 142
Completed | 128 | 139
Not Completed | 14 | 3
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Various reasons | 8 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ioforminol 320mg I/ml Injection | Iopamidol 370mg I/ml Injection | Total
Number analyzed (Participants) | 137 | 141 | 278
Age, Categorical [Count of Participants; unit: Participants] — Per a Protocol Amendment, A-01, the minimum age changed to male or female greater than or equal to 18 years of age who have a history of chronic renal insufficiently.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 28 | 30 | 58
    >=65 years | 109 | 111 | 220
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 53 | 101
  Male | 89 | 88 | 177
Region of Enrollment [Number; unit: participants]
  United States | 128 | 134 | 262
  Canada | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Overall Image Quality Between Ioforminol and Iopamidol-enhanced Images as Determined by an Independent Reader.
Description: Overall image quality (excellent, adequate or poor) and diagnostic usefulness (diagnostic or non-diagnostic) were assessed using qualitative scales.
Time Frame: After the imaging date for either Ioforminol or Iopamidol.
Population: The measured values are looking at 1) Overall Image Quality and, 2) Diagnostic Usefulness.
Measure: Number; unit: Number of subjects
Arm/Group | Ioforminol 320mg I/ml Injection | Iopamidol 370mg I/ml Injection
Number analyzed (Participants) | 137 | 141
Number of subjects
  Overall Image Quality-Excellent | 65 | 71
  Overall Image Quality-Adequate | 57 | 59
  Overal Image Quality-Poor | 15 | 11
  Diagnostic Usefulness-Diagnostic | 123 | 134
  Diagnostic Usefulness-Non-Diagnostic | 14 | 7

2. Secondary Outcome: To Determine Incidence Rates of the Overall AEs, Organ-specific AEs (i.e., Delayed Skin Reactions, General Subject Comfort, and Allergic/Immunologic Reactions, Etc.) and SAEs Following Administration
Description: To determine incidence rates of the overall AEs, organ-specific AEs (i.e., delayed skin reactions, general subject comfort, and allergic/immunologic reactions, etc.) and SAEs following administration of GE-145 or iopamidol.
  To determine incidence rates and onset time of biomarker-based and SCr-based CI-AKI following administration of GE-145 or iopamidol.
  Summary of Treatment-Emergent Adverse Events (TEAE) in greater than of equal to 2% of Subjects.
Time Frame: Time zero equals the date of contrast imaging and for up to 7 days for safety monitoring post contrast administration.
Population: Summary of Treatment-Emergent Adverse Events (TEAE) in greater than of equal to 2% of Subjects.
Measure: Number; unit: Number of events
Arm/Group | Ioforminol 320mg I/ml Injection | Iopamidol 370mg I/ml Injection
Number analyzed (Participants) | 137 | 141
Number of events
  Angina Pectoris | 3 | 2
  Coronary Artery Disease | 3 | 3
  Diarrhea | 3 | 1
  Nausea | 3 | 3
  Catheter-Site Hematoma | 9 | 8
  Catheter-Site Hemorrhage | 4 | 6
  Catheter-Site Pain | 4 | 3
  Chest Pain | 3 | 2
  Urinary Tract Infection | 3 | 4
  Blood Creatinine Increased | 2 | 4
  Pain In Extremity | 2 | 5
  Dizziness | 0 | 3
  Headache | 11 | 1

3. Secondary Outcome: Assessing the Incidence of Renal Biomarker-based Contrast-induced Acute Kidney Injury (CI-AKI) in Subjects Post Administration of Ioforminol or Iopamidol Injections
Description: Analyzing the number of subjects with renal biomarker-based contrast-induced acute kidney injury (CI-AKI).
Time Frame: 2, 6 and 24 hours post Ioforminol and Iopamidol adminstration
Population: Summary of subjects with renal biomarker-based CI-AKI by time point (Per Protocol Population).
Measure: Number; unit: Subjects
Arm/Group | Ioforminol 320mg I/ml Injection | Iopamidol 370mg I/ml Injection
Number analyzed (Participants) | 109 | 106
Subjects
  Time- Post Contrast, 2 hours | 24 | 21
  Time- Post Contrast, 6 hours | 48 | 33
  Time- Post Contrast, 24 hourss | 61 | 49

ADVERSE EVENTS:
Time Frame: Up to 7 days post Ioforminol and Iopamidol administrations.
Groups:
- Ioforminol 320mg I/ml Injection: Ioforminol 320 mg I/mL as a single iv. administration. Up to 7 days post Iopamidol administration.
- Iopamidol 370mg I/ml Injection: Iopamidol 370 mg I/mL as a single iv. administration. Up to 7 days post Ioforminol administration.
Arm/Group | Ioforminol 320mg I/ml Injection | Iopamidol 370mg I/ml Injection
Serious Adverse Events (participants affected / at risk) | 13/137 | 10/141
Other Adverse Events (participants affected / at risk) | 20/137 | 9/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ioforminol 320mg I/ml Injection (N=137) | Iopamidol 370mg I/ml Injection (N=141)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
Aortic stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Congestive cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (2)
Coronary artery disease and hospitalization (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Unstable angina (Cardiac disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Vascular pseudoaneurysm to hospitalization (General disorders) | 1 (1) | 0 (0)
Dyspnea (General disorders) | 0 (0) | 1 (1)
Hematoma (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Coronary artery bypass (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac pacemaker insertion to hospitalization (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ioforminol 320mg I/ml Injection (N=137) | Iopamidol 370mg I/ml Injection (N=141)
Catheter-Site Hemotoma (General disorders) | 9 (9) | 8 (8) — Site of Administration
Headache (Nervous system disorders) | 11 (11) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No